CLINICAL TRIAL: NCT04977232
Title: Game Intervention as Adjunct Therapy for Anhedonia in Patients With Major Depressive Disorder
Brief Title: Adjunctive Game Intervention for Anhedonia in MDD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Guo Wenbin, Professor of Psychiatry Department of Psychiatry of the Second Xiangya Hospital, Central South University, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYG2021038
Record Dates: First submitted 2021-07-13; First posted 2021-07-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Escitalopram + game intervention (Experimental): Escitalopram treatment and game intervention are given in combinations for 8 weeks.
  Interventions: Drug: Escitalopram; Behavioral: Game intervention
- Escitalopram (Active Comparator): Escitalopram treatment for 8 weeks
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Selective serotonin reuptake inhibitors (SSRI) were most commonly used first line pharmacotherapy for depression.
  Other Names: Lexapro
Behavioral: Game intervention — Participants will be instructed to play the commercial video game for about 30-60 minutes at least three times per week.
  Arms: Escitalopram + game intervention

SUMMARY:
This is a pilot study using game intervention as an adjuvant treatment, to evaluate the effect of the video game on anhedonia and associated functional change of brain in patients with depression. Participants will be randomized to Experimental group receiving a 8-week treatment of antidepressant drugs and game intervention, or Control group receiving a 8-week treatment of antidepressant drugs. Magnetic resonance imaging scanning and assessment of clinical characteristics and cognitive function were conducted before and after the intervention.

DETAILED DESCRIPTION:
Depression is a serious mental health problem that affects millions of people globally. Anhedonia, a core symptom of depression, is the loss of pleasure or interest in enjoyable activities. The presence of anhedonia is a risk factor of poor outcome of depression. Although some patients reach remission after treatment, anhedonia still persists as a residual symptom. It is generally believed that the frontal-striatal pathway plays an important role in the reward system of brain in patients with depression. The mechanism of anhedonia is closely related to the function of the brain's reward system dopamine. There have been some research showed benefits of playing video games on brain. Video games can modulate negative emotions and increase positive feelings. Previous studies have confirmed that playing games will activate the release of dopamine in striatum. "Dancing Line" is a commercial music game. Participants need to change the direction of target according to the music by tapping the screen and manage to finish the routes and get the gems along the route as much as possible. Sometimes the view of participants would change during the game. The game is simple for participants to pick up and there is no need for prior gaming experience. The main purpose of the study is to explore the effect of game as an adjuvant treatment on anhedonia, depressive symptoms, cognitive function and associated functional change of brain in patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of Major Depressive Disorder according to DSM IV or V and validated via Mini International Neuropsychiatric Interview (M.I.N.I.)
* right handedness
* capability of understanding and finishing self-rating scales
* capability of providing informed consent

Exclusion Criteria:

* any other major psychiatric disorders following DSM-5 diagnostic criteria
* neurological diseases
* a history of drug abuse
* suicidal risk
* pregnancy
* any contraindication for brain MRI scan.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Snaith-Hamilton-Pleasure Scale (SHAPES) | From baseline to 8 weeks
  Pre-post assessment of anhedonia via the Snaith-Hamilton-Pleasure Scale (SHAPES). Raw score range is 14-56. A higher score indicates a worse outcome.
Temporal Experience of Pleasure Scale (TEPS) | From baseline to 8 weeks
  Pre-post assessment of anhedonia via the Temporal Experience of Pleasure Scale (TEPS). Raw score range is 20-120. A lower score indicates a worse outcome.
Hamilton Depression Rating scale (HAMD) | From baseline to 8 weeks
  Pre-post assessment of depressive symptoms via Hamilton Depression Rating scale (HAMD). Raw score range is 0-52. Higher scores indicate more severe depression.

SECONDARY OUTCOMES:
Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | From baseline to 8 weeks
  Pre-post assessment of cognitive function via Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).
The Stroop test | From baseline to 8 weeks
  Pre-post assessment of cognitive function via the Stroop test.
Wisconsin Card Sorting Test (WCST) | From baseline to 8 weeks
  Pre-post assessment of cognitive function via Wisconsin Card Sorting Test (WCST).
Rumination Responses Scale | From baseline to 8 weeks
  Pre-post assessment of rumination via Rumination Responses Scale. Raw score range is 22-88. Higher scores indicate worse outcomes.
Magnetic Resonance Imaging data | From baseline to 8 weeks
  Whole brain Magnetic Resonance Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Guo, Principal Investigator — Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, China